CLINICAL TRIAL: NCT01565772
Title: A Phase I Trial of Hypofractionated Proton Radiation Therapy With Cisplatin and Etoposide Followed by Surgery in Stage III Non-Small Cell Lung Cancer
Brief Title: Proton Radiation Therapy With Cisplatin and Etoposide Followed by Surgery in Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Henning Willers, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-253
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung cancer; Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Proton Therapy; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation, Chemotherapy and Surgery (Experimental): Proton beam radiation, plus chemotherapy with cisplatin and etoposide, followed by surgery.
  Interventions: Radiation: Proton Beam Radiation; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Radiation: Proton Beam Radiation — 45-55 Gy total, 1.8-2.2 Gy x 25 fractions Mon-Fri for 5 weeks
Drug: Cisplatin — 50 mg/m2 IV on days 1, 8 of cycles 1 and 2
Drug: Etoposide — 50 mg/m2 IV on days 1-5 on Cycles 1-2

SUMMARY:
This research study is looking at an alternative way of delivering radiation therapy with protons. Protons are tiny particles with a positive charge that can be controlled to travel a certain distance and stop inside the body. In theory, this allows better control of where the radiation dose is delivered as compared to photons. Information from other research studies suggests that proton radiation may help to reduce unwanted side effects from radiation and allow an increase in radiation dose that increase the odds of tumor killing.

The purpose of this study is to determine the safest dose of proton radiation therapy to give in combination with standard chemotherapy in participants with Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Proton radiation will be delivered daily Monday through Friday for 5 weeks. Study therapy will be give as an outpatient at the Francis H. Burr Proton Center at Massachusetts General Hospital.

During the weeks that subjects receive radiation, they will also receive 2 cycles of chemotherapy. Each cycle will last 28 days.

Cisplatin will be give as an IV infusion over 30-60 minutes or 1-2 hours on Days 1 and 8 of Cycles 1 and 2.

Etoposide will be given as an IV infusion over 60 minutes on Days 1, 2, 3, 4, 5 of Cycles 1 and 2.

After radiation and 2 cycles of chemotherapy are completed, subjects may have surgery to remove their tumor.

Following surgery, subjects may receive another 2 cycles of chemotherapy (Cycles 3 and 4). Each cycles lasts 21 days. Cisplatin is given on Day 1. Etoposide is given on Days 1, 2, and 3.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer with a clinical stage of IIIA
* Candidate for chemoradiation and surgical resection
* Measurable disease
* Life expectancy > 6 months
* Normal organ and marrow function

Exclusion Criteria:

* Pregnant or breast-feeding
* Prior therapy for lung cancer with chemotherapy
* Prior chest radiation
* Compromised pulmonary function
* Severe neurovascular disease
* History of high cardiac risk including unstable angina
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin or etoposide
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive hear failure, unstable angina pectoris, clinically significant or serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of a different malignancy unless disease-free for at least 3 years and at low risk for recurrence. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, non muscle-invasive bladder cancer, basal cell or squamous cell carcinoma of the skin
* Subjects with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
MTD | 1.5 years
  To establish the MTD of a proton beam-based regimen consisting of 25 fractions, together with concurrent standard cisplatin and etoposide chemotherapy followed by surgery +/- adjuvant chemotherapy for Stage III NSCLC, and to describe post-treatment surgical complications and treatment toxicity using CTCAE v4.0

SECONDARY OUTCOMES:
Downstaging and Response | 1.5 years
  To describe pathological downstaging and response following preoperative proton radiation and cisplatin/etoposide chemotherapy
Biomarkers | 1.5 years
  To explore the predicitive value of biomarkers for radio- and chemosensitization in pre-treatment tumor biopsies and surgical specimens.
Tumor Control and Survival Rates | 5 years
  To evaluate local and regional tumor control rates, progression free survival (PFS) rates, and overall survival rates and 2 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henning Willers, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States